CLINICAL TRIAL: NCT05137327
Title: Examining Outcomes of a Multi-Component, Individually-Tailored Consultation Process Focused on Classroom Management for Teachers
Brief Title: Classroom Behavior Support (CBS) Project
Acronym: CBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Julie Owens, Professor of Psychology, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-F-16; R324A190154 (Other Grant/Funding Number: Institute of Education Sciences)
Record Dates: First submitted 2021-11-28; First posted 2021-11-30 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-12

CONDITIONS: ADHD
Keywords: inattention; disruptive behavior
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Problem Behavior | interventions — Cystathionine beta-Synthase

STUDY DESIGN:
Intervention Model Description: Within a given school building, teachers will be stratified on three characteristics prior to randomization: (1) grade bands (K-2 and 3-5), (2) Global Classroom Management Competencies based on baseline observations and (3) teacher beliefs based on baseline ratings. This will ensure that similar numbers of teachers with these characteristics are in each condition.
Who Masked: Participant
Masking Description: Teachers are unaware of the consultation condition to which they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classroom Behavior Support (CBS) Condition (Experimental): Consultants follow the problem-solving process used in the comparison condition and attempt to address barriers to integrity using the knowledge, skills, beliefs, or stress components in the CBS manual. Consultants conduct a Values Interview, so teacher values can be used in the individual goal setting and decision making process. Consultants are trained to (a) incorporate the teacher's values into the problem-solving process, (b) elicit change talk from teachers using techniques borrowed from Motivational Interviewing, and (c) engage in Socratic questioning and cognitive restructuring for beliefs that may be barriers to integrity (e.g., "should" statements). Enhanced performance feedback involves highlighting connections between teacher integrity and child outcomes and using this as a catalyst for a knowledge, skills, beliefs, or stress component. Consultants use change rulers to elicit motivation to achieve the stated goals.
  Interventions: Behavioral: Classroom Behavior Support (CBS) Condition
- Standard Problem Solving Comparison Condition (Active Comparator): Consultation in the comparison condition follows a 5-step problem solving approach and provide brief performance feedback procedures that mirror (in duration, content, and process) best practice procedures (Gilbertson et al., 2007; Noell et al., 1997). The guiding principles for this condition are that the performance feedback portion of the session should be limited to 5 to 10 minutes and unless the teacher initiates discussion of other content, the problem solving should remain student-focused, rather than teacher-focused. Discussion on teacher values and beliefs, and attempts to facilitate change talk, are contra-indicated. If the teacher initiates discussion of knowledge, beliefs, or skills, the consultant may answer questions, but may not use strategies associated with Motivational Interview or Cognitive-Behavioral Therapy (CBT) or strategies in CBS condition. We have separate scripts and checklists for each condition.
  Interventions: Behavioral: Standard Problem Solving Consultation

INTERVENTIONS:
Behavioral: Classroom Behavior Support (CBS) Condition — An individualized teacher consultation program that includes observation and performance feedback and techniques borrowed from Motivational Interviewing and Cognitive Behavioral Therapy (CBS). It is designed to address barriers to implementation and improve teacher practices and student outcomes.
  Arms: Classroom Behavior Support (CBS) Condition
Behavioral: Standard Problem Solving Consultation — A standard problem solving approach to teacher consultation that includes observation and brief performance feedback. It represents current best practice in teacher consultation.
  Arms: Standard Problem Solving Comparison Condition

SUMMARY:
The goal of the study is to conduct a randomized clinical trial to evaluate the impact of the Classroom Behavior Support Program (CBS; a multi-component, individually-tailored teacher consultation program) on teachers' classroom management practices (universal and targeted) and resulting student behavioral and educational outcomes relative to a best practices comparison consultation condition.

DETAILED DESCRIPTION:
Participants will be 165 general education teachers (teaching Kindergarten through 6th grade) who have room for growth in classroom management skills, along with their classroom of students and one target student with inattentive and/or disruptive behavior problems. Teachers will be recruited over 3 cohorts (1 cohort per year). Teachers will be randomly assigned to one of two consultation conditions and participate for an entire academic year. Teachers in both conditions will be scheduled to receive consultation every other week between August and December and one time per month between January and March. The focus of the consultation will be teacher implementation of universal classroom management practices (Tier 1) and the targeted intervention applied with the target student (either a daily report card and organization intervention; Tier 2). Teachers will be observed weekly and data from observation will be incorporated into consultation sessions. Investigators will examine the main effects of consultation on growth in teacher practices (universal and targeted) and change in proximal and distal student outcomes (classwide and in target students), as well as the mediators and moderators of these effects.

ELIGIBILITY:
Inclusion Criteria:

TEACHER INCLUSION CRITERIA:

Teacher of a general education class in a participating elementary school (teacher grades K-6th grade) with at least one of the following from observation screening data.

* Below 51% response to student rule violations;
* A rate of praise per hour that falls below the 30th percentile for teachers of the same grade;
* A rate of student rule violations that exceeds the 70th percentile for that grade.

STUDENT INCLUSION CRITERIA:

* Student must spend at least 50% of his/her day in the teacher's classroom
* Student must receive at three or more scores that are lower than a 3 on a positive Daily Behavior Rating (DBR) subscale or three or more scores higher than 3 on a negative DBR subscale.
* Parents must provide consent.

Exclusion Criteria:

TEACHER: no exclusionary criteria.

STUDENT: Special education eligibility of cognitive disability, autism, or multiple disability.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Teacher Percent Appropriate Response to Rule Violation (ARRV) - Whole Class (Tier 1 Teacher Outcome) | Growth from baseline through study completion, an average of 8 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, each student rule violation is tallied using a frequency count procedure. Following each rule violation, teacher responses are coded. Investigators calculate a percent appropriate response for each observation. Scores range from 0% to 100%; higher scores represent better response. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Teacher Percent Appropriate Response to Rule Violation (ARRV) - Target Student (Tier 2 Teacher Outcome) | Growth from baseline through study completion, an average of 6 months
  Once the target student is identified and consented (typically 2 months after the start of school), target student behaviors are observed using the Using the Student Behavior-Teacher Response (SBTR) observation system. Each target student rule violation is tallied using a frequency count procedure. Following each rule violation, teacher responses are coded. Investigators calculate a percent appropriate response for each observation. Scores range from 0% to 100%; higher scores represent better response. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Whole Class Student Rule Violations (Tier 1 Student Outcome) | Change from baseline through study completion, an average of 8 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, each student rule violation is tallied using a frequency count procedure. Using the observation duration, investigators calculate a rate per hour. Scores range from 0 to any upper limit; higher numbers represent more classwide rule violations per hour. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Target Student Rule Violations (Tier 2 Student Outcome) | Change from baseline through study completion, an average of 6 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, target student rule violations are tallied using a frequency count procedure. Using the observation duration, investigators calculate a rate per hour. Scores range from 0 to any upper limit; higher numbers represent more target student rule violations per hour. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.

SECONDARY OUTCOMES:
Teacher Rate of Praise - Whole Class (Tier 1 Teacher Outcome) | Change from baseline through study completion, an average of 8 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, each instance of praise (labeled and unlabeled) is tallied using a frequency count procedure. Using the observation duration, investigators calculate a rate of praise per hour. Scores range from 0 to any upper limit; higher numbers represent more teacher praise statements per hour. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Teacher Rate of Praise - Target Student (Tier 2 Teacher Outcome) | Change from baseline through study completion, an average of 6 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, each instance of praise (labeled and unlabeled) directed at the target student is tallied using a frequency count procedure. Using the observation duration, investigators calculate a rate of praise per hour. Scores range from 0 to any upper limit; higher numbers represent more teacher praise statements made to the target student per hour. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Teacher Rate of Opportunities to Respond (OTR) - Whole Class (Tier 1 Teacher Outcome) | Change from baseline through study completion, an average of 8 months
  Using the Student Behavior-Teacher Response (SBTR) observation system, each Opportunity to Respond (OTR; a question asked to a group of children that facilitates engaged attention) is tallied using a frequency count procedure. Using the observation duration, investigators calculate a rate of OTRs per hour. Scores range from 0 to any upper limit; higher numbers represent more teacher use of OTRs per hour. Observations are conducted weekly for the duration of the trial (30-minutes each). Data are averaged across observations between consultation sessions.
Teacher Ratings of Target Student Academic Performance - (Tier 2 Student Outcome) | Growth from baseline through study completion, an average of 6 months
  Teachers complete the Academic Performance Rating Scale (APRS) on target students at baseline and on a monthly basis following the launch of the Tier 2 intervention. The APRS is a 19-item scale comprised of two subscales assessing children's' Academic Success (i.e., academic achievement) and Academic Productivity (i.e., day-to-day performance).
Teacher Ratings of Target Student Behavior - (Tier 2 Student Outcome) | Change from baseline through study completion, an average of 6 months
  Teachers complete the Strengths and Difficulties Questionnaire (SDQ) on target students at baseline and on a monthly basis following the launch of the Tier 2 . The SDQ is a 25 item behavioral screening questionnaire that includes subscales assessing conduct problems and hyperactivity/inattention. Items on each subscale range from 0 to 10; higher scores indicate more problematic behaviors.
Parent Ratings of Target Student Behavior - (Tier 2 Student Outcome) | Change from baseline to study completion, an average of 6 months
  Parents complete the Strengths and Difficulties Questionnaire (SDQ) on target students at baseline and at the end of the school year (fall and spring). The SDQ is a 25 item behavioral screening questionnaire that includes subscales assessing conduct problems and hyperactivity/inattention. Items on each subscale range from 0 to 10; higher scores indicate more problematic behaviors.
Teacher Ratings of Target Student ADHD Symptoms - (Tier 2 Student Outcome) | Change from baseline to study completion, an average of 6 months
  Teachers complete the ADHD Rating Scale-5 at baseline and at the end of the school year (fall and spring). The ADHD Rating Scale-5 assess the symptoms of ADHD as described in the DSM-5 (9 symptoms of inattention; 9 symptoms of Hyperactivity-Impulsivity) and associated impairments in functioning. Scores for each subscale range from 0 to 27; higher scores indicate more severe symptoms in that domain.
Parent Ratings of Target Student ADHD Symptoms - (Tier 2 Student Outcome) | Change from baseline to study completion, an average of 6 months
  Parent complete the ADHD Rating Scale-5 at baseline and at the end of the school year (fall and spring). The ADHD Rating Scale-5 assess the symptoms of ADHD as described in the DSM-5 (9 symptoms of inattention; 9 symptoms of Hyperactivity-Impulsivity) and associated impairments in functioning. Scores for each subscale range from 0 to 27; higher scores indicate more severe symptoms in that domain.
Teacher Ratings of Positive and Problematic Student Behaviors - (Tier 2 Student Outcome) | Change from baseline to study completion, an average of 6 months
  Teachers complete four, 5-item Daily Behavior Ratings (DBR) on target students at baseline and on a monthly basis following the launch of the Tier 2 intervention. Teachers rate positive behaviors in two domains: Organizational Skills (5 items) and Engagement (5 items) and problem behaviors in two domains: Oppositional (5 items), and Disruptive (5 items) behavior. Scores range from 0 to 35. Higher scores on the positive domains indicate better organization skills and engagement. Higher scores on the negative domains indicate more sever problems in each area.
Target Student Grade Point Average (GPA) Intervention Year - (Tier 2 Student Outcome) | Growth from baseline to study completion, an average of 6 months
  Investigators will collect quarterly grades during the intervention year and calculate a 4-point GPA using core academic subjects. Scores range from 0 to 4; higher scores indicate better academic achievement.
Target Student Grade Point Average (GPA) Long Term Follow Up - (Tier 2 Student Outcome) | Growth from baseline to one year following study completion, an average of 18 months
  Among students whose parents given consent for us to track their child's GPA in the year following intervention, investigators will collect quarterly grades during the year following the intervention year and calculate a 4-point GPA using core academic subjects. Scores range from 0 to 4; higher scores indicate better academic achievement.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Within one year of end of the project period, the final project data will be fully de-identified and stored in SPSS files with accompanying documents that describe the variables, the measures, and the project procedures.
  We will post on our center's web pages that data requests for this study can be made online. Instructions for submitting such requests will be clearly described on the web pages. All requests, related correspondence, and outcome of the requests will be stored in our center.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This will become available 1 year after the end of the study and will be available for 10 years after we publish the main findings of the study.
Access Criteria: Receiving parties must (a) identify the primary contact person and multiple means of contact, (b) identify any other persons who will have access to the data, (c) specify the research questions and the nature of the analyses, and confirm that the contact person/s has the expertise to use the data to achieve those goals, (d) specify the planned outlet for the findings, and (e) sign an agreement that (1) they will maintain the dataset in a private and confidential location, not share the data with any parties outside those specified in (a) and (b), and not manipulate the data for the purposes of attempting to identify participants, and (2) they will give Drs. Owens and Evans the opportunity to review and comment on any product prior to dissemination, and give them the opportunity to be a co-author on the product if desired.
URL: http://www.oucirs.org